CLINICAL TRIAL: NCT03539744
Title: A Phase 3, Multicenter, Randomized, Open Label Study of Venetoclax and Dexamethasone Compared With Pomalidomide and Dexamethasone in Subjects With t(11;14)-Positive Relapsed or Refractory Multiple Myeloma
Brief Title: A Study Designed to Evaluate the Safety and Efficacy of Venetoclax Plus Dexamethasone (VenDex) Compared With Pomalidomide Plus Dexamethasone (PomDex) in Participants With t(11;14)-Positive Relapsed or Refractory Multiple Myeloma.
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M13-494; 2023-506112-40 (Other: EU CT)
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2018-05-17; First posted 2018-05-29 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
Keywords: Cancer, Multiple Myeloma (MM), Relapsed or Refractory Multiple Myeloma (R/R MM), pharmacokinetics; CANOVA
MeSH Terms: conditions — Multiple Myeloma; Neoplasms; Recurrence | interventions — pomalidomide; Dexamethasone; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 VenDex (Experimental): Venetoclax administered orally once daily (QD) plus dexamethasone administered orally once every week (Q1W) for each 28-day cycle.
  Interventions: Drug: Dexamethasone; Drug: Venetoclax
- Arm 2 PomDex (Active Comparator): Pomalidomide administered orally once daily (QD) on Days 1 - 21 for each 28-day cycle plus dexamethasone administered orally once every week (Q1W) for each 28-day cycle.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pomalidomide — capsule, oral
  Other Names: Pomalyst
  Arms: Arm 2 PomDex
Drug: Dexamethasone — oral, locally available form
Drug: Venetoclax — tablet; oral
  Other Names: ABT-199; GDC-0199
  Arms: Arm 1 VenDex

SUMMARY:
A study designed tocompare progression-free survival (PFS) in participants with t(11;14)-positive MM treated with venetoclax in combination with dexamethasone versus pomalidomide in combination with dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of multiple myeloma (MM) based on standard International Myeloma Working Group (IMWG) criteria.
* Measurable disease at screening as defined per protocol.
* Has received at least 2 prior lines of therapy as described in the protocol.
* Has had documented disease progression on or within 60 days after completion of the last therapy.
* Has received at least 2 consecutive cycles of lenalidomide and be relapsed/refractory to lenalidomide, as defined per protocol.
* Has received at least 2 consecutive cycles of a proteasome inhibitor (PI).
* Has t(11;14)-positive status determined by an analytically validated fluorescent in situ hybridization (FISH) assay per centralized laboratory testing.
* An Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Laboratory values (liver, kidney and hematology laboratory values) that meet criteria as described per protocol.

Exclusion Criteria:

* History of treatment with venetoclax or another B-Cell Lymphoma (BCL)-2 inhibitor or pomalidomide.
* History of other active malignancies, including myelodysplastic syndromes (MDS), within the past 3 years (exceptions described in the protocol).
* Evidence of ongoing graft-versus-host disease (GvHD) if prior stem cell transplant (SCT).
* Prior treatment with any of the following: allogeneic or syngeneic SCT within 16 weeks prior to randomization; or autologous SCT within 12 weeks prior to randomization.
* Known central nervous system involvement of MM.
* Concurrent conditions as listed in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 43 months from first randomization
  PFS is defined as the time in days from subject randomization to the date of the first documented progressive disease (PD) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 43 months from first randomization
  ORR is defined as the percentage of participants with documented best response (sCR, CR, VGPR or partial response [PR]) prior to first documented PD.
Very Good Partial Response or Better Response Rate (VGPR) | Up to approximately 43 months from first randomization
  VGPR or better response rate is defined as the proportion of participants with documented stringent complete response (sCR), complete response (CR), or VGPR.
Overall survival (OS) | Up to approximately 51 months from first randomization
  OS is defined as the number of days from the date that the participant was randomized to the date of the participant's death.
Minimal Residual Disease (MRD) Negativity Rate | Up to approximately 43 months from first randomization
  MRD defined as the percentage of participants with MRD negativity status. MRD negativity will be defined at 10^-5 threshold as measured by centralized testing of bone marrow aspirate samples by next generation sequencing (NGS).
Time to Deterioration in Disease Symptoms | Up to approximately 51 months from first randomization
  Time to deterioration in disease symptoms is measured by the disease symptom domain of the European Organization for Research and Treatment of Cancer Quality of Life Multiple Myeloma Module 20 (EORTC QLQ-MY20).
Time to Deterioration in Physical Functioning | Up to approximately 51 months from first randomization
  Time to deterioration in physical functioning is measured by the physical functioning domain of European Organization for Research and Treatment of Cancer Quality of Life Core 30 Question Questionnaire (EORTC-QLQ-C30).
Change from Baseline in PROMIS Fatigue Score | Up to approximately 51 months from first randomization
  Change from baseline in the Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form 7a score.
Change from Baseline in BPI-SF Worst Pain Score | Up to approximately 51 months from first randomization
  Change from baseline in the Brief Pain Inventory - Short Form (BPI-SF) worst pain score.
Change from Baseline in EuroQoL 5 Dimension 5 Level (EQ-5D-5L) | Up to approximately 51 months from first randomization
  EQ-5D-5L consists of 2 components: the EQ-5D descriptive system and the EQ visual analog scale (VAS). The EQ-5D descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS records the participant's self-rated health on a vertical VAS where the endpoints are labelled "The best health you can imagine" and "The worst health you can imagine."
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Up to approximately 51 months from first randomization
  EORTC QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including 5 functional scales (physical, role, emotional, social, and cognitive), 3 symptom scales (fatigue, nausea and vomiting, and pain), a global health status/quality of life scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties).
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Multiple Myeloma Module 20 (EORTC QLQ-MY20) | Up to approximately 51 months from first randomization
  EORTC QLQ-MY20 includes scales for disease symptoms, side effects of treatment, future perspective, and body image. Values for each scale range from 0 to 100.
Duration of response (DOR) | Up to approximately 43 months from first randomization
  DOR for a participant is defined as the number of days from the date of first documented response (PR or better) to the date of first documented PD or death due to multiple myeloma, whichever occurs first.
Time to Disease Progression (TTP) | Up to approximately 43 months from first randomization
  TTP for a participant is defined as the number of days from the date of randomization to the date of first documented PD or death due to multiple myeloma, whichever occurs first.
Time to Response (TTR) | Up to approximately 43 months from first randomization
  TTR for a participant is defined as the number of days from the date of randomization to the date of first documented response (PR or better).
Cmax of Venetoclax | Up to approximately 225 days from initial dose
  Maximum plasma concentration (Cmax) of venetoclax
Trough Concentration (Ctrough) of Venetoclax | Up to approximately 225 days from initial dose
  Observed plasma concentration at trough (Ctrough) of venetoclax.
Number of Participants With Adverse Events (AEs) | Up to approximately 51 months from first randomization
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (180):
- United States (19):
  - Duplicate_University of Arizona Cancer Center - North Campus /ID# 218407, Tucson, Arizona
  - VA Central California Health Care System /ID# 200047, Fresno, California
  - University of California, Los Angeles /ID# 171524, Los Angeles, California
  - Rocky Mountain Regional VA Medical Center/Eastern Colorado Health Care System /ID# 222904, Aurora, Colorado
  - Mayo Clinic /ID# 200075, Jacksonville, Florida
  - Cleveland Clinic Florida /ID# 208884, Weston, Florida
  - Duplicate_Norton Cancer Institute /ID# 200834, Louisville, Kentucky
  - University of Maryland, Baltimore /ID# 217422, Baltimore, Maryland
  - Boston Medical Center /ID# 223606, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer In /ID# 201377, Detroit, Michigan
  - Duplicate_Henry Ford Hospital /ID# 171531, Detroit, Michigan
  - Mayo Clinic - Rochester /ID# 201091, Rochester, Minnesota
  - Columbia University Medical Center /ID# 200715, New York, New York
  - Fairview Hospital - Moll Pavilion /ID# 208919, Cleveland, Ohio
  - Cleveland Clinic Main Campus /ID# 202247, Cleveland, Ohio
  - UPMC Hillman Cancer Ctr /ID# 200063, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center at Texas Medical Center /ID# 200060, Houston, Texas
  - Huntsman Cancer Institute /ID# 218406, Salt Lake City, Utah
  - VA Puget Sound Health Care System /ID# 222708, Seattle, Washington
- Australia (7):
  - Liverpool Hospital /ID# 202431, Liverpool, New South Wales
  - Sydney Adventist Hospital /ID# 222874, Wahroonga, New South Wales
  - Wollongong Hospital /ID# 205545, Wollongong, New South Wales
  - ICON Cancer Care - Townsville /ID# 206565, Hyde Park, Queensland
  - Icon Cancer Centre /ID# 205663, South Brisbane, Queensland
  - The Queen Elizabeth Hospital /ID# 202432, Woodville South, South Australia
  - Perth Blood Institute Ltd /ID# 206649, Nedlands, Western Australia
- Canada (4):
  - Arthur J. E. Child Comprehensive Cancer Centre /ID# 218846, Calgary, Alberta
  - BC Cancer - Vancouver /ID# 222804, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre - Victoria General /ID# 218883, Halifax, Nova Scotia
  - CISSS-CA (Centre Integre de sante et de services sociaux de Chaudiere-Appalache) /ID# 218887, Lévis, Quebec
- China (21):
  - Beijing Chaoyang Hospital,Capital Medical University /ID# 216014, Beijing, Beijing Municipality
  - Peking University Third Hospital /ID# 216371, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital (East) - Dongdan Campus /ID# 216040, Beijing, Beijing Municipality
  - Sun Yat-Sen University Cancer Center /ID# 223828, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital /ID# 215860, Guangzhou, Guangdong
  - Henan Cancer Hospital /ID# 215987, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 215850, Wuhan, Hubei
  - Nanjing Drum Tower Hospital /ID# 223143, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University /ID# 216094, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 216954, Nanchang, Jiangxi
  - The First Hospital of China Medical University /ID# 215996, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University /ID# 223435, Shenyang, Liaoning
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 216643, Shanghai, Shanghai Municipality
  - Shanghai Tongji Hospital /ID# 218865, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University /ID# 216647, Chengdu, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sc /ID# 216041, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital /ID# 223550, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 215989, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 218691, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University /ID# 218953, Wenzhou, Zhejiang
  - Beijing Chaoyang Hospital, Capital Medical University(West campus) /ID# 234033, Beijing
- Czechia (5):
  - Fakultní Nemocnice Brno - Jihlavská /ID# 204512, Brno, Brno-mesto
  - Fakultní nemocnice Hradec Králové - Sokolská /ID# 221291, Hradec Králové, Hradec Kralove
  - Fakultni Nemocnice Ostrava /ID# 204515, Ostrava, Ostrava-mesto
  - Fakultni nemocnice Olomouc /ID# 221290, Olomouc
  - Vseobecna fakultni nemocnice v Praze /ID# 221166, Prague
- Denmark (5):
  - Duplicate_Herlev Hospital /ID# 223221, Herlev, Capital Region
  - Aalborg University Hospital /ID# 223220, Aalborg, North Denmark
  - Odense University Hospital /ID# 223217, Odense, Region Syddanmark
  - Sygehus Lillebalt, Vejle /ID# 223216, Vejle, Region Syddanmark
  - Duplicate_Roskilde Hospital /ID# 223366, Roskilde
- France (10):
  - Duplicate_CHU Grenoble - Hopital Michallon /ID# 223182, La Tronche, Isere
  - CHU Reims - Hôpital Robert Debre /ID# 233907, Reims, Marne
  - CHRU Nancy - Hopitaux de Brabois /ID# 201076, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHRU Lille - Hopital Claude Huriez /ID# 202213, Lille, Nord
  - Hopitaux Universitaires Henri Mondor - Hopital Henri Mondor /ID# 202211, Créteil, Paris
  - CHU de Nantes, Hotel Dieu -HME /ID# 200099, Nantes, Pays de la Loire Region
  - HCL - Hopital Lyon Sud /ID# 200097, Pierre-Bénite, Rhone
  - Centre Henri Becquerel /ID# 223186, Rouen, Seine-Maritime
  - CH Henri Duffaut /ID# 234154, Avignon, Vaucluse
  - Hopital Pitie Salpetriere /ID# 214173, Paris, Île-de-France Region
- Germany (9):
  - Robert-Bosch-Krankenhaus /ID# 223947, Stuttgart, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen /ID# 238646, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Wuerzburg /ID# 200055, Würzburg, Bavaria
  - Klinikum Chemnitz gGmbH /ID# 233797, Chemnitz, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 201830, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Jena /ID# 201254, Jena, Thuringia
  - Charite Universitaetsklinikum Berlin - Campus Benjamin Franklin /ID# 200051, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 215495, Hamburg
  - Asklepios Klinik Altona /ID# 222506, Hamburg
- Greece (6):
  - Alexandra General Hospital /ID# 202386, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 222879, Heraklion, Crete
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 213982, Athens
  - University Gen Hosp of Patra /ID# 201691, Pátrai
  - Theageneio Anticancer Hospital /ID# 213983, Thessaloniki
  - General Hospital of Thessaloniki George Papanikolaou /ID# 201692, Thessaloniki
- Israel (9):
  - Rambam Health Care Campus /ID# 169678, Haifa, H_efa
  - Bnai Zion Medical Center /ID# 169466, Haifa, H_efa
  - The Lady Davis Carmel Medical Center /ID# 222969, Haifa, H_efa
  - Hadassah /ID# 169474, Jerusalem, Jerusalem
  - Duplicate_Assuta Ashdod Medical Center /ID# 222968, Ashdod, Southern District
  - Soroka University Medical Center /ID# 218768, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 169778, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 169437, Tel Aviv, Tel Aviv
  - Rabin Medical Center /ID# 244611, Petah Tikva
- Italy (7):
  - Duplicate_IRCCS AOU di Bologna - Policlinico Sant'Orsola-Malpighi /ID# 170952, Bologna, Emilia-Romagna
  - A.O.U. CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO - Ospedale Molinette /ID# 170962, Turin, Piedmont
  - Irccs-Crob /Id# 170955, Rionero in Vulture, Potenza
  - Azienda Ospedaliero Universitaria delle Marche /ID# 170950, Ancona
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 212498, Milan
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello /ID# 222988, Palermo
  - Azienda Ospedaliera Santa Maria Terni /ID# 170948, Terni
- Japan (18):
  - Nagoya City University Hospital /ID# 170880, Nagoya, Aichi-ken
  - The Jikei University Kashiwa Hospital /ID# 223031, Kashiwa-shi, Chiba
  - Kyushu University Hospital /ID# 171117, Fukuoka, Fukuoka
  - Ogaki Municipal Hospital /ID# 171043, Ogaki-shi, Gifu
  - Gunma University Hospital /ID# 170966, Maebashi, Gunma
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital /ID# 171255, Hiroshima, Hiroshima
  - Kobe City Medical Center General Hospital /ID# 170992, Kobe, Hyōgo
  - Duplicate_National Hospital Organization Mito Medical Center /ID# 171187, Higashi Ibaraki-gun, Ibaraki
  - Hitachi General Hospital /ID# 200843, Hitachi-shi, Ibaraki
  - Iwate Medical University Hospital /ID# 222849, Shiwa-gun, Iwate
  - Tohoku University Hospital /ID# 201935, Sendai, Miyagi
  - Okayama Medical Center /ID# 200119, Okayama, Okayama-ken
  - Japanese Red Cross Osaka Hospital /ID# 171493, Osaka, Osaka
  - The University of Osaka Hospital /ID# 201966, Suita-shi, Osaka
  - Tokushima University Hospital /ID# 202571, Tokushima, Tokushima
  - The Jikei University Hospital /ID# 239014, Minato-ku, Tokyo
  - Japanese Red Cross Medical Center /ID# 171256, Shibuya-ku, Tokyo
  - Yamagata University Hospital /ID# 238329, Yamagata, Yamagata
- Russia (7):
  - Moscow State budget healthcare /ID# 169685, Moscow, Moscow
  - Research Institute of Fundamental and Clinical Immunology /ID# 223594, Novosibirsk, Novosibirsk Oblast
  - LLC Novaya Klinika /ID# 169689, Pyatigorsk, Stavropol Kray
  - City Clinical Hospital #52 /ID# 206289, Moscow
  - Leningrad Regional Clinical Hospital /ID# 202776, Saint Petersburg
  - Almazov National Medical Research Centre /ID# 169681, Saint Petersburg
  - Tula Regional Clinical Hospital /ID# 223226, Tula
- Singapore (3):
  - National University Hospital /ID# 203988, Singapore
  - Singapore General Hospital /ID# 202131, Singapore
  - Tan Tock Seng Hospital /ID# 204374, Singapore
- South Korea (6):
  - Duplicate_Gachon University Gil Medical Center /ID# 202827, Incheon, Gyeonggido
  - Seoul National University Hospital /ID# 202711, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 202710, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 234045, Seoul, Seoul Teugbyeolsi
  - Ulsan University Hospital /ID# 222716, Ulsan, Ulsan Gwang Yeogsi
  - Yonsei University Health System Severance Hospital /ID# 202709, Seoul
- Spain (14):
  - Hospital Universitari Son Espases /ID# 222889, Palma de Mallorca, Balearic Islands
  - Hospital Costa del Sol /ID# 234083, Marbella, Malaga
  - Complejo Hospitalario Universitario Ourense /ID# 222876, Ourense, Ourense
  - Hospital Universitario Canarias /ID# 238452, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Universitario Vall d'Hebron /ID# 218106, Barcelona
  - Instituto Catalan de Oncologia (ICO) Girona /ID# 171311, Girona
  - Hospital de Leon /ID# 233878, León
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 171304, Madrid
  - Disc_Hospital Universitario 12 de Octubre /ID# 171288, Madrid
  - Hospital Universitario La Paz /ID# 218107, Madrid
  - Hospital Universitario de Salamanca /ID# 171294, Salamanca
  - Hospital Universitario Virgen del Rocio /ID# 171286, Seville
  - Hospital General Universitario de Toledo /ID# 222887, Toledo
  - Hospital Universitario y Politecnico La Fe /ID# 234019, Valencia
- Sweden (4):
  - Sunderby sjukhus /ID# 201314, Luleå, Norrbotten County
  - Sodra Alvsborgs sjukhus /ID# 213061, Borås, Västra Götaland County
  - Duplicate_Universitetssjukhuset Linköping /ID# 200789, Linkoping, Västra Götaland County
  - Uddevalla sjukhus /ID# 201315, Uddevalla, Västra Götaland County
- Turkey (Türkiye) (9):
  - Cukurova Universitesi Tip Fakultesi /ID# 201955, Saricam Adana, Adana
  - Izmir Ekonomi Universitesi Ozel Medicalpoint Hastanesi /ID# 201954, Cordaleo, İzmir
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi /ID# 201956, Ankara
  - Gazi University Medical Faculty /ID# 222698, Ankara
  - Ankara Univ Medical Faculty /ID# 201881, Ankara
  - Istanbul University Istanbul Medical Faculty /ID# 201953, Istanbul
  - Bagcilar Medipol Mega Universite Hastanesi /ID# 222914, Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi /ID# 201952, Istanbul
  - Ege University Medical Faculty /ID# 222697, Izmir
- Ukraine (5):
  - Communal Nonprofit Enterprise Cherkasy Regional Oncology Dispensary /ID# 223943, Cherkasy, Cherkasy Oblast
  - Communal non-profit enterprise Regional Center of Oncology /ID# 223945, Kharkiv, Kharkivs’ka Oblast’
  - MNI Khmelnytskyi Regional Hospital of Khmelnytskyi Regional Council /ID# 223942, Khmelnytskyi
  - National Cancer Institute /ID# 223944, Kyiv
  - SI Institute of Blood Pathology and Transfusion Medicine of NAMS of Ukraine /ID# 223941, Lviv
- United Kingdom (12):
  - Addenbrooke's Hospital /ID# 223097, Cambridge, Cambridgeshire
  - Hammersmith Hospital /ID# 171446, London, England
  - University College London Hospital /ID# 171428, London, Greater London
  - Norfolk and Norwich University Hospitals NHS Foundation Trust /ID# 218213, Norwich, Norfolk
  - Duplicate_Nottingham University Hospitals NHS Trust /ID# 223292, Nottingham, Nottinghamshire
  - Duplicate_NHS Greater Glasgow and Clyde /ID# 202199, Glasgow, Scotland
  - Duplicate_University Hospitals North Midlands - Royal Stoke University Hospital /ID# 218355, Stoke-on-Trent, Staffordshire
  - Duplicate_Duplicate_Lewisham and Greenwich NHS Trust /ID# 171445, London
  - Manchester University NHS Foundation Trust /ID# 171440, Manchester
  - Portsmouth Hospitals University NHS Trust /ID# 171444, Portsmouth
  - Royal Berkshire NHS Foundation Trust /ID# 217835, Reading
  - Duplicate_Sheffield Teaching Hospitals NHS Foundation Trust - Royal Hallamshire /ID# 171447, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Popat R, Beksac M, Dimopoulos MA, Gatt ME, Gay F, Jo JC, Kapoor P, Katodritou E, Kortum KM, Ling S, Nagarajan C, Suzuki K, Qiu L, Onishi M, Ku G, Dail M, Mukherjee N, Ross JA, Badawi MA, Fusco MJ, Dobkowska E, Arriola E, Bueno OF, Bahlis NJ, Iida S, Moreau P, Valent J, Mateos MV. Venetoclax-Dexamethasone Versus Pomalidomide-Dexamethasone in t(11;14)-Positive Relapsed/Refractory Multiple Myeloma: Primary Results of the Randomized, Phase III CANOVA Study. J Clin Oncol. 2026 Jan 20;44(3):164-175. doi: 10.1200/JCO-25-00924. Epub 2025 Dec 10. PMID 41370738
- See also: Related info — https://www.abbvieclinicaltrials.com/study/?